CLINICAL TRIAL: NCT06597045
Title: BIOMARKER and IMAGING CHARACTERISATION of INFLAMMATORY ATHEROMA in PATIENTS RECEIVING IMMUNOTHERAPY and ANGIOGENESIS INHIBITORS
Acronym: BIOCAPRI
Status: Active, not recruiting | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Roche Diagnostics GmbH (Industry); University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: INGN21CA318
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer; Cardiotoxicity; Atherosclerotic Disease
Keywords: cancer; atherosclerosis; FDG; PETCT; cardiotoxicity; VEGFI; immune checkpoint inhibitor
MeSH Terms: conditions — Neoplasms; Cardiotoxicity; Atherosclerosis | interventions — Positron Emission Tomography Computed Tomography; Blood Specimen Collection; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine biomarkers will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Immune checkpoint inhibitor monotherapy: Patients who are given immune checkpoint inhibitor (ICI) monotherapy (decision on treatment is made by the clinical oncology team. Enrolment to this study had no influence or impact on choice of anti-cancer therapy.
  Patients were allocated this group if they received at least one cycle of immune check point inhibitor. In the event that a patient is given ICI/VEGFI combination therapy but the VEGFi was stopped early (due to toxicity or lack of clinical effect, determined by the clinical team) and they had less than 50% exposure to VEGFi in the protocol window (24 weeks), the patient will be allocated to ICI monotherapy. Subsequent sensitivity analyses looking at any exposure to VEGFI vs those who had no exposure will be performed.
  Interventions: Diagnostic Test: PET/CT with 18-FDG
- VEGF inhibitor monotherapy: Patients who are given VEGF inhibitor monotherapy (decision on treatment is made by the clinical oncology team. Enrolment to this study had no influence or impact on choice of anti-cancer therapy
  Patients will be allocated this group if they are given VEGFi with no exposure to immunotherapy in the study period. If patients are enrolled in the study but stop VEGF inhibitor early they will still be included in this group, provided they do not receive immune checkpoint inhibitor. If during the study protocol window, the patient is exposed to other anti-cancer therapies (other than ICI), in addition to VEGF inhibitor, they will be remain in the VEGFI group.
  Interventions: Diagnostic Test: PET/CT with 18-FDG
- Immune checkpoint inhibitor / VEGF inhibitor combination therapy: Patients who are given immune checkpoint inhibitor / VEGF inhibitor combination therapy (decision on treatment is made by the clinical oncology team. Enrolment to this study had no influence or impact on choice of anti-cancer therapy).
  Patients were allocated this group if they received at least one cycle of immune check point inhibitor and VEGFI with more than 50% of the exposure in the study protocol window (24 weeks). Subsequent sensitivity analyses looking at any exposure to VEGFI vs those who had no exposure will be performed.
  Interventions: Diagnostic Test: PET/CT with 18-FDG

INTERVENTIONS:
Diagnostic Test: PET/CT with 18-FDG — Study specific tests will include 18F-FDG PET/CT (specialised CT scan), electrocardiography (ECG), clinic blood pressure assessment, blood tests, urine sample, echocardiography (heart ultrasound) and tests on the fingertips (EndoPAT).
  Positron emission tomography with computerised tomography (PET-CT) is a scanning technique in routine clinical use. It is the gold standard method for assessing blood vessel inflammation. A small amount of radioactive sugar (18F-FDG [18F- fluorodeoxyglucose]) is administered intravenously 90 minutes prior to the PET-CT scan. The distribution of uptake of this tracer is seen on the subsequent PET-CT scan. The CT component of this scan allows the PET image to be precisely aligned with anatomical structures (especially large blood vessels).
  Other Names: blood and urine biomarkers; endopat; echocardiography

SUMMARY:
The advent of immunotherapy (immune checkpoint inhibitors [ICI]) has been an extremely important advancement for cancer treatment in recent decades. The anti-cancer effects of these agents is profound and can lead to radiological 'disappearance' of the primary cancer and metastatic deposits. ICI are now commonly used in the treatment of multiple cancers including melanoma, kidney cancer, liver cancer and lung cancer. ICI can be used on their own or in combination with other agents such as vascular endothelial growth factor inhibitors (VEGFi) which is first line treatment for many patients. However, it has become clear that these drugs have cardiovascular side effects including high blood pressure and a reduction in the heart muscle pumping function. It is also increasingly recognised that ICIs may have a toxic effect on blood vessels resulting in an increased risk of heart attack or stroke. These side effects can have a significant impact on patients' health and can lead to withdrawal of important cancer treatment. The mechanisms by which these side effects occur are unclear and have not been well described to date.

The aim of this study is to examine the effect of ICI and VEGFi, both alone and in combination, on blood vessels and to understand their effects on blood markers and heart function. This study is observational and will not require any modification of cancer therapy.

This study will aim to recruit patients diagnosed with cancer who are already planned to receive ICI or VEGFi alone or in combination at the Beatson West of Scotland Oncology Centre. Patients will undergo a vascular PET-CT scan before and 6 months after starting treatment. In addition patients will undergo echocardiography and tests of the function of the small blood vessels in the fingertips with a special machine (EndoPat). Blood and urine samples will also be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cancer who are planned for treatment with ICI or VEGFI, including combination therapy
2. ≥6 months predicted survival
3. Age ≥18 years

Exclusion Criteria:

1. Patients who are unable or unwilling to provide valid consent for the study
2. Patients with diabetes who are on oral anti-diabetic treatment or insulin at baseline
3. patients who have exposure to either immune checkpoint inhibitor or VEGF inhibitor in the 12 months before enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending oncology clinics at the the Beatson West of Scotland Oncology Centre with a diagnosis of cancer and planned for treatment with ICI and/or VEGFi therapies will be screened for entry into the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-10-14 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Mean arterial TBRmax 18F FDG uptake | 24 weeks
  Inflammatory plaque activity (meanMaxTBR)* in patients receiving ICI/VEGFI combination therapy versus ICI alone or VEGFI alone.
  *Note 'meanMaxTBR' is a PET measurement reflecting the average of the maximum 'target to background ratio [TBR]) where 'target' denotes regions of PET radiotracer activity)

SECONDARY OUTCOMES:
Blood and urine biomarker analysis | Baseline (pre-treatment) to 24 weeks
  Correlation between baseline and longitudinal changes in humoral/urinary biomarkers as potential predictors of subsequent change in inflammatory plaque activity (TBR).
  Analysis of blood and urine biomarkers with inflammatory plaque activity (meanMaxTBR) in patients receiving ICI (alone or in combination) vs VEGFI alone.
Inflammatory plaque activity (meanMaxTBR) in patients receiving ICI (alone or in combination) vs VEGFI alone. | Baseline (pre-treatment) to 24 weeks
  In addition to ICI vs VEGFI vs ICI/VEGFI combination therapy, we will also compare PET activity in those who had ICI (monotherapy or combination therapy) with VEGFi monotherapy.
PET activity with baseline cardiovascular risk factors and imaging (echo/CT) | Baseline (pre-treatment) to 24 weeks
  Correlation between baseline cardiovascular risk factors and imaging (echo/CT) findings will be examined as predictors of subsequent change in inflammatory plaque activity (TBR).
The effect of ICI/VEGFI upon endothelial function (EndoPAT) will be examined. | Baseline (pre-treatment) to 24 weeks
  The effect of ICI/VEGFI upon endothelial function (EndoPAT) will be examined.
PETCT 18F FDG uptake arterial analyses | Baseline (pre-treatment) to 24 weeks
  In accordance with European Association of Nuclear Medicine guidelines, in addition to TBRmax, arteries will be analysed using TBRmean (tissue to background ratio mean FDG uptake), active segment; and most diseased segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom